CLINICAL TRIAL: NCT03485235
Title: Effect of Dilatation and Curettage on the Endometrial Receptivity and Pregnancy Outcome in Patients With Recurrent Implantation Failure
Brief Title: Effect of Dilatation and Curettage on the Endometrial Receptivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed S Sweed, MD, Principal Investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AS1764
Record Dates: First submitted 2018-03-26; First posted 2018-04-02 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Embryo Implantation
MeSH Terms: interventions — Sperm Injections, Intracytoplasmic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- D&C (Experimental)
  Interventions: Procedure: D&C; Procedure: ICSI
- No D&C (Other)
  Interventions: Procedure: ICSI

INTERVENTIONS:
Procedure: D&C — Dilatation and curettage
  Arms: D&C
Procedure: ICSI — Intra Cytoplasmic Sperm Injection

SUMMARY:
Effect of dilatation and curettage on the endometrial receptivity and pregnancy outcome in patients with recurrent implantation failure

ELIGIBILITY:
Inclusion Criteria:

1. All the patients had at least 3 failed trials of IVF-ET with day 5 fresh blastocyst transferred
2. At least 10 high-grade embryos were obtained in the previous trials
3. Level of AMH more than or equal 1.1 ng/ml.
4. Age: Less than or equal to 35 years

Exclusion Criteria:

1. Patients with uterine pathology e.g. myoma , Asherman syndrome, Septum ,adenomyosis
2. Hydrosalpinx
3. Endometriosis
4. patients with diagnosed autoimmune diseases affecting pregnancy e.g. S.L.E.

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2018-03-31 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-12-10 (Actual)

PRIMARY OUTCOMES:
Live Birth Rate | 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Maternity Hospital, Cairo, Egypt